CLINICAL TRIAL: NCT02709590
Title: Randomized Clinical Trial of Oral Diclofenac Potassium With Cervical Lidocaine Cream in Reducing Pain During HSG
Brief Title: Diclofenac Potassium With Lidocaine Cream in Reducing Pain During HSG
Acronym: DP-L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HS3
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Pain Relief With HSG
MeSH Terms: interventions — Diclofenac; Lidocaine; Psychotherapy, Multiple

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): oral diclofenac potassium plus lidocaine anesthetic cream placed into their cervix immediately before HSG
  Interventions: Drug: diclofenac potassium + lidocaine
- Group B (Placebo Comparator): oral placebo tablets plus placebo cream placed into their cervix immediately before HSG
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: diclofenac potassium + lidocaine — patients will have of oral diclofenac potassium 60 minutes before the procedure plus lidocaine anesthetic cream placed into their cervix immediately before HSG
  Other Names: combined therapy
  Arms: Group A
Drug: placebo — patients will have of oral placebo tablet 60 minutes before the procedure plus placebo cream placed into their cervix immediately before HSG
  Arms: Group B

SUMMARY:
The aim of our study is to determine the efficacy of oral diclofenac potassium combined with lidocaine cream on the pain scores during HSG.

ELIGIBILITY:
Inclusion Criteria:

* any patient came for HSG

Exclusion Criteria:

* any patient has contraindication to HSG

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean pain score during hysterosalpigography by visual analog scale | intraoperative

SECONDARY OUTCOMES:
Mean pain score after hysterosalpigography | 30 minutes
side effects of medication | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided